CLINICAL TRIAL: NCT02103972
Title: Assessment of Efficacy of the Consumption of a Heat-treated Lactobacillus Paracasei (GM080) on Atopic Dermatitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 11.46.NRC
Record Dates: First submitted 2014-03-26; First posted 2014-04-04 (Estimated); Last update posted 2018-01-26 (Actual); Status verified 2018-01

CONDITIONS: Atopic Dermatitis
Keywords: All subjects of any ethnicity aged from 4 to 30 months with atopic dermatitis skin symptoms with a SCORAD equal or above 20
MeSH Terms: conditions — Dermatitis, Atopic | interventions — maltodextrin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Maltodextrin (Placebo Comparator): Maltodextrin
  Interventions: Dietary Supplement: Maltodextrin
- GM080 (Active Comparator): GM080
  Interventions: Dietary Supplement: GM080

INTERVENTIONS:
Dietary Supplement: GM080
  Arms: GM080
Dietary Supplement: Maltodextrin
  Arms: Maltodextrin

SUMMARY:
The primary objective of this trial is to assess the efficacy of the consumption of heat-treated Lactobacillus paracasei (GM080) on atopic dermatitis as compared to a placebo treatment.

ELIGIBILITY:
Inclusion Criteria:

* Infants aged from 4-30 months (inclusive) at the time of enrolment (63 in each group).
* With mild to severe atopic symptoms: SCORAD ≥ 20 (at V0b).
* Having obtained his/her (or his/her legal representative's) written Informed Consent.

Exclusion Criteria:

* SCORAD inferior to 20 (SCORAD less than 20 at V0b). A SCORAD less than 20 at V0c is not an exclusion criteria.
* Infants who need a systemic treatment for their skin condition (e.g. glucocorticoids, steroids, cyclosporine A).
* Infants or mothers who introduce probiotics (other than the study product) in their diet during the 16-weeks intervention study. Of note: Infants or mothers who are used to consume a certain probiotic for more than 1 month before the start of the study (V0b), can continue to use this probiotic during the intervention period and will not be excluded. Recent introduction of probiotics, within a month before the planned start of the study (V0b) should be stopped and recorded; at least 1 month should be between stopping the consumption of the probiotic and V0b).
* Infants having other inflammatory skin diseases (urticaria, psoriasis).
* Infants having a congenital illness or malformation that may affect normal growth (especially immunodeficiency).
* Infants whose parents/caregivers cannot be expected to comply with the study procedures.
* Infants currently participating or having participated in another clinical study during the last 4 weeks prior to the beginning of this study.
* Infants using topical calcineurin inhibitors (e.g. tacrolimus and pimecrolimus (ELIDEL®)) during the study.
* Infants who have undergone in the month before the start of the study (V0b), are currently undergoing or are anticipated to undergo ultraviolet light therapy or wet dressing or any other topical treatment of their eczema other than the one provided in the study. Lotion and skin moisturizer are allowed but need to be monitored for frequency and area.
* The investigator and clinician will assess if the child has to be excluded based on the patient's medical condition and taken into account the values of the safety parameters tested. Therefore, no cut-off values, or normal ranges for the different safety parameters are exclusion criteria. It will be the responsibility of the investigator and clinician, based on their medical judgement, to decide if it is safe or not to include an infant into the study.

Ages: 4 Months to 30 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 126 (Actual)
Dates: Start 2014-07; Primary Completion 2017-07 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
Change from Baseline SCORAD Score at 16 weeks of treatment | between 0 and 16 weeks of treatment
  SCORAD documented during the longitudinal observational period of 16 weeks after the subject has enrolled

SECONDARY OUTCOMES:
Score A, B and C of the SCORAD | 0, 4, 10 and 16 weeks of treatment
  Score A, B and C of the SCORAD The scores A, B and C of the SCORAD as well as the subcategories of the scores B and C will be analyzed separately (measured at V0c, V1, V2 and V3)
Number and duration of atopic dermatitis episodes | during the 16 weeks intervention period
  Number and duration of atopic dermatitis episodes The number of episodes of atopic dermatitis and the total number of days with symptoms during the 16 weeks intervention period
Transepidermal water loss | 0, 4, 10 and 16 weeks
  TEWL will be measured at V0, V1, V2 and V3 on 4 sites of both non-lesional and lesional appearing skin parts
Topical treatment used | during the 16 weeks of treatment
  Topical treatment used (sparing effect) The corticoid sparing effect of the ingredient will be assessed in the placebo and the ingredient group.
total and specific IgE | 0 and 16 weeks
  total and specific IgE
Quality of Life | 0, 4, 10, 16 weeks and 1 and 4 years later
  The infants' dermatitis quality of life index (IDQOL) will be collected
assess the effect of the product on the safety parameters | 0 and 16 weeks
  Biochemistry and Hematology parameters
"Objective" SCORAD, which is composed of part A and B of the SCORAD (measured at V0, V1, V2 and V3) | 0, 4, 10 and 16 weeks

OTHER OUTCOMES:
Diaper rash episodes and duration will be recorded by the parents/caregivers | duting the 16 weeks of treatment
  Diaper rash episodes and duration will be recorded by the parents/caregivers
Perception/impression of the ingredient by the caregiver | at 16 weeks
  At the end of the 16 weeks intervention trial, the perception of the caregivers toward the ingredient they were randomized to, will be assessed
Assessment of allergic history and skin disease | 1 and 4 years later
Cytokine quantification | 0 and 16 weeks of treatment
  Cytokine quantification (multiplex) will be assessed in plasma of the patients
Genetic characterization of atopic dermatitis associated polymorphism | 0 week
  Five major mutations in the FLG gene, one polymorphism in SPINK5 and one insertion in KLK7 gene will be analyzed in blood DNA

CONTACTS AND LOCATIONS:
Locations (6):
- Taiwan (6):
  - Kaohsiung Municipal TA-TUNG Hospital, Kaohsiung City, Qianjin District
  - Kaohsiung Municipal Hsiao-Kang Hospital, Kaohsiung City, Siaogang District
  - Taipei Chang Gung Memorial Hospital of the Chang-Gung Medical foundation, Taipei, Songshan District
  - Chung Shan Medical University Hospital, Taichung, South District
  - Linkou Chang Gung Memorial Hospital, Gueishan Township, Taoyuan County
  - Cardinal Tien Hospital, New Taipei City, Xindian District